CLINICAL TRIAL: NCT00901329
Title: NEXGEN Gender Fixed Bearing Knee Versus NEXGEN LPS-Flex Fixed Bearing Knee - a Prospective Randomized Study Comparing Two Different Knee Prostheses
Brief Title: NexGen Gender Fixed Bearing Knee Versus NexGen Legacy Knee Posterior Stabilized (LPS) - Flex Fixed Bearing Knee: A Study Comparing Two Different Knee Prostheses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Henrik Husted, Orthopedic department, Hvidovre University Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD2007-0123
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Total Knee Arthroplasty
Keywords: TKA; functional outcome; pain; ROM; gait
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Gender prosthesis (Experimental)
  Interventions: Device: NexGen Gender Fixed Bearing Knee prosthesis
- 2: LPS flex prosthesis (Active Comparator)
  Interventions: Device: NexGen LPS-Flex Fixed Bearing Knee prosthesis

INTERVENTIONS:
Device: NexGen Gender Fixed Bearing Knee prosthesis — new female prosthesis
  Arms: 1: Gender prosthesis
Device: NexGen LPS-Flex Fixed Bearing Knee prosthesis — standard knee prosthesis
  Arms: 2: LPS flex prosthesis

SUMMARY:
The purpose of this trial is to study potential differences between two prostheses, including: "feel of prosthesis" (i.e., how natural does the prosthesis feel), range of motion (ROM), pain perception for each prosthesis, satisfaction, patella tracking and quantification of the removed bone anterior on the femur (weight).

DETAILED DESCRIPTION:
The present study compares the Gender prosthesis against the LPS-flex in a bilateral study, where patients are given two different prostheses: Gender on one side and LPS-flex on the other side. Patients are blinded to which prosthesis is selected for which side. The potential advantages of the Gender prosthesis include: less post-op pain due to better sizing (less overhang), less post-op patellofemoral pain and less compromised extensor mechanism and better patella tracking (due to less overstuffing of the patellofemoral joint).

Design:

The study is prospective, randomized, comparative and blinded. 24 female patients scheduled for simultaneous bilateral total knee arthroplasty are included (48 knees).

Power calculations cannot be performed as to how many patients are needed since no previous studies have been conducted.

All patients are included and operated by consultant Henrik Husted.

Methods:

Patients are randomized to which side is operated with which prosthesis (LPS-flex or Gender); the operations are performed using standard instrumentation and standard approaches.

At the operation the weight of the cut bone from the anterior femur is noted for each side. Before discharge radiographs including skyline views are performed to evaluate patella tracking (and are repeated at the final out-patient check 1 year post-op).

Gait analyses are performed before operation and 1 year post-op. All other procedures are standard procedures already implemented in the department.

Patients follow an accelerated track (ANORAK, 1,2) with an intended LOS of 4 days for bilaterally operated knee-arthroplasties, all patients are discharged directly to their homes.

ELIGIBILITY:
Inclusion Criteria:

* female patients scheduled for simultaneous bilateral total knee arthroplasty (TKA) are included
* bilateral knee disease necessitating bilateral TKA

Exclusion Criteria:

* male sex

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
follow-up at 6 weeks, 3 months, 6 months and one year. - knee-score and function score - feel of prosthesis (VAS 0-10) - ROM (max passive and active ROM is measured using a goniometer) - pain (VAS 0-10) - satisfaction (VAS 0-10) | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Hvidovre, Copenhagen
  - orthopedic department, section of arthroplasty, Hvidovre University Hospital, Copenhagen, Hvidovre